CLINICAL TRIAL: NCT07271524
Title: Investigation of the Plasticity of Deep Brain Structures in Mild Cognitive Impairment and Healthy Aging (PlasMA)
Brief Title: Non-invasive Deep Brain Stimulation to Improve Spatial Navigation Abilities in Individuals Following Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friedhelm Hummel (Other)
Collaborators: Fondation Bertarelli (Unknown); The Novartis Foundation (Other); Clinique Romande de Readaptation (Network); HUG University hospital (Unknown); SNF Swiss National Foundation (Unknown); Wyss Center for Bio and Neuroengineering (Other); Fondation Akiva (Unknown); Canton du Valais (Unknown)
Responsible Party: Sponsor-Investigator, Friedhelm Hummel, Professor, Defitech Chair of Clinical Neuroengineering Brain Mind Institute, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-00127-wp73t; 2020-00127 (Other: Commission cantonale d'Éthique de la Recherche sur l'être humain Vaud (CER-VD))
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
Keywords: non-invasive brain stimulation; deep brain stimulation; subcortical; memory; neuro-imaging; transcranial temporal interference stimulation; spatial navigation; electroencephalography; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Spatial Navigation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Patterned stimulation (intermittent theta-burst) generating temporal interference in the hippocampal-entorhinal complex; see Beanato et al. 2024, Sci Adv (DOI: 10.1126/sciadv.ado4103) for details.
  Interventions: Other: Transcranial electric stimulation
- Control stimulation (Placebo Comparator): High-frequency (2kHz) electrical stimulation with no frequency shift, generating no temporal interference.
  Interventions: Other: Transcranial electric stimulation

INTERVENTIONS:
Other: Transcranial electric stimulation — Transcranial temporal interference stimulation (tTIS) is an innovative non-invasive brain stimulation approach, in which two or more independent stimulation channels deliver high-frequency currents in the kHz range (oscillating at f1 and f1 + Δf). These high-frequency currents are assumed to be too high to effectively modulate neuronal activity. Still, by applying a small shift in frequency, they result in a modulated electric field with the envelope oscillating at the low-frequency Δf (target frequency) where the two currents overlap. The peak of the modulated envelope amplitude can be steered towards specific areas located deep in the brain, by tuning the positions of the electrodes and the current ratio across stimulation channels. Here, the investigators apply tTIS via surface electrodes applying a low-intensity, sub-threshold protocol following the safety guidelines for low-intensity transcranial electric stimulation in humans.

SUMMARY:
Impairments in spatial memory and spatial navigation are commonly reported amongst patients presenting post-traumatic brain injury (TBI). In this study, the investigators examine the effect of non-invasive deep brain stimulation of the hippocampal-entorhinal complex (HC-EC), a key region supporting navigation abilities, on spatial navigation performance in TBI patients. Using a virtual reality task where participants must first encode and later recall the location of objects in a virtual arena, the investigators contrast performance while active versus control stimulation is applied to the HC-EC. The investigators additionally record brain activity using electroencephalography (EEG) prior to, during, and after task performance to characterize the neural correlates of spatial navigation abilities in TBI patients, and how they are affected by stimulation.

DETAILED DESCRIPTION:
Patients will perform a virtual reality spatial navigation task comparable to that used previously by Beanato and colleagues (2024; DOI: 10.1126/sciadv.ado4103). Patients will perform 4 blocks of task, each lasting approximately 10 minutes; during the full duration of each block, either active or control transcranial temporal interference stimulation (tTIS) will be applied in an interleaved manner, and EEG recordings will be collected. Resting-state EEG recordings will also be collected prior to and following task performance.

Structural, diffusion-weighted, and resting-state MRI scans will additionally be performed during a prior baseline session.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of TBI
* No history of other severe neurological or psychiatric disorders

Exclusion Criteria:

* Unable to consent
* Severe neuropsychiatric (e.g., major depression, severe dementia) or unstable systemic diseases (e.g., severe progressive and unstable cancer, life threatening infectious diseases)
* Severe sensory or cognitive impairment or musculoskeletal dysfunctions prohibiting to understand instructions or to perform the experimental tasks
* Inability to follow or non-compliance with the procedures of the study
* Contraindications for NIBS or MRI:

  * Electronic or ferromagnetic medical implants/device, non-MRI compatible metal implant
  * History of seizures
  * Medication that significantly interacts with NIBS being benzodiazepines, tricyclic antidepressants and antipsychotics
* Regular use of narcotic drugs
* Pregnancy
* Request of not being informed in case of incidental findings
* Concomitant participation in another trial involving probing of neuronal plasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Speed in the spatial navigation task | During intervention (approximate duration of intervention = 40 minutes, administered in a single session)
  Participant speed (in seconds) of departure to, and reach of, object location in the virtual reality spatial navigation task.
Accuracy in the spatial navigation task | During intervention (approximate duration of intervention = 40 minutes, administered in a single session)
  Accuracy (error, in virtual meters, between correct and recalled object location) in the virtual reality spatial navigation task.

SECONDARY OUTCOMES:
Brain oscillatory activity | Peri-interventional (up to 1 hour; approximate duration of intervention = 40 minutes, administered in a single session)
  Resting-state and task-related EEG recordings are collected, and metrics of oscillatory activity are extracted to characterize the neural activity associated to the primary outcome.
Brain structure and connectivity | Baseline (before the intervention)
  Structural, diffusion-weighted, and resting-state MRI scans are performed during the baseline session and are used to evaluate inter-individual anatomical factors associated to the primary outcome.

OTHER OUTCOMES:
Age (years) | Baseline (before the intervention)
  Participant age will be recorded to examine its influence on individual responsiveness to the intervention.
Montreal Cognitive Assessment questionnaire score | Baseline (before the intervention)
  Participant score on the Montreal Cognitive Assessment questionnaire will be collected to examine its influence on individual responsiveness to the intervention.
Frontal Assessment Battery questionnaire score | Baseline (before the intervention)
  Participant score in the Frontal Assessment Battery questionnaire will be collected to examine its influence on individual responsiveness to the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - EPFL, Campus Biotech, Geneva, Canton of Geneva
  - EPFL Valais, Clinique Romande de readaptation, Sion, Valais

IPD SHARING:
Plan to Share IPD: Undecided